CLINICAL TRIAL: NCT02645682
Title: The Effects of Anti-infective Central Venous Catheter(CVC) on Catheter-related Bloodstream Infection(CRBSI) in Critical Care Patients: a Multiple-center, Randomized, Control Study
Brief Title: The Effects of Anti-infective Central Venous Catheter on Catheter-related Infection in Critically Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Kang Yan, professor; chief physician, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HC-I-H 1503
Record Dates: First submitted 2015-12-30; First posted 2016-01-05 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Critical Illness
Keywords: central venous catheter (CVC); catheter-related bloodstream infection (CRBSI); catheter-related thrombosis (CRT)
MeSH Terms: conditions — Critical Illness

ARMS (2):
- anti-infection CVC (Certofix®protect) (Experimental): intervention group
  Interventions: Device: anti-infection CVC
- normal CVC (Certofix®) (Active Comparator): control group
  Interventions: Device: normal CVC

INTERVENTIONS:
Device: anti-infection CVC
  Other Names: Certofix®protect
  Arms: anti-infection CVC (Certofix®protect)
Device: normal CVC
  Other Names: Certofix®
  Arms: normal CVC (Certofix®)

SUMMARY:
The purpose of this study is to investigate the effect of anti-infective central venous catheter(Certofix®Protect) on reducing catheter-related bloodstream infection in critically ill patients in China, and the relationship between catheter-related bloodstream infection and catheter-related thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* adult patients in intensive care unit (ICU)（age ≥ 18 years）
* needs double lumen CVC more than 5 days
* Signed informed consent

Exclusion Criteria:

* thrombosis in target and/or contralateral vein
* pregnancy or lactating women
* unlikely to survive for more than 1 month
* bad prognosis
* suspected catheter-related infection
* replacement CVC in original site through guide wire
* severe burn
* situation that is not suitable for CVC, including allergic to CVC material, thrombosis in target vein, infection of puncture site, coagulation disorder, abnormal anatomy
* already in this study
* participated in other studies within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1818 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
catheter-related bloodstream infection | through study completion, an average of 2 years
  number of participants with catheter-related bloodstream infection

SECONDARY OUTCOMES:
catheter-related thrombosis | through study completion, an average of 2 years
  number of participants with catheter-related thrombosis
all cause mortality | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yan Kang, Doctor, Study Chair — West China Hospital; Bin Du, Doctor, Study Chair — Peking Union Medical College Hospital
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan

REFERENCES:
- [Background] O'Grady NP, Alexander M, Burns LA, Dellinger EP, Garland J, Heard SO, Lipsett PA, Masur H, Mermel LA, Pearson ML, Raad II, Randolph AG, Rupp ME, Saint S; Healthcare Infection Control Practices Advisory Committee. Guidelines for the prevention of intravascular catheter-related infections. Am J Infect Control. 2011 May;39(4 Suppl 1):S1-34. doi: 10.1016/j.ajic.2011.01.003. No abstract available. PMID 21511081
- [Background] Cicalini S, Palmieri F, Petrosillo N. Clinical review: new technologies for prevention of intravascular catheter-related infections. Crit Care. 2004 Jun;8(3):157-62. doi: 10.1186/cc2380. Epub 2003 Sep 29. PMID 15153233
- [Background] Saint S, Veenstra DL, Lipsky BA. The clinical and economic consequences of nosocomial central venous catheter-related infection: are antimicrobial catheters useful? Infect Control Hosp Epidemiol. 2000 Jun;21(6):375-80. doi: 10.1086/501776. PMID 10879567
- [Background] 中华医学会重症医学分会。血管内导管相关感染的预防与治疗指南。中国实用外科杂志2008; 28: 413-21
- [Background] Rupp ME. Central venous catheters coated or impregnated with antimicrobial agents effectively prevent microbial colonisation and catheter-related bloodstream infections. Evid Based Med. 2014 Apr;19(2):56. doi: 10.1136/eb-2013-101471. Epub 2013 Sep 5. No abstract available. PMID 24009330
- [Background] Halton KA, Cook DA, Whitby M, Paterson DL, Graves N. Cost effectiveness of antimicrobial catheters in the intensive care unit: addressing uncertainty in the decision. Crit Care. 2009;13(2):R35. doi: 10.1186/cc7744. Epub 2009 Mar 11. PMID 19284570
- [Background] Maki DG, Stolz SM, Wheeler S, Mermel LA. Prevention of central venous catheter-related bloodstream infection by use of an antiseptic-impregnated catheter. A randomized, controlled trial. Ann Intern Med. 1997 Aug 15;127(4):257-66. doi: 10.7326/0003-4819-127-4-199708150-00001. PMID 9265424
- [Background] Raad I, Darouiche R, Dupuis J, Abi-Said D, Gabrielli A, Hachem R, Wall M, Harris R, Jones J, Buzaid A, Robertson C, Shenaq S, Curling P, Burke T, Ericsson C. Central venous catheters coated with minocycline and rifampin for the prevention of catheter-related colonization and bloodstream infections. A randomized, double-blind trial. The Texas Medical Center Catheter Study Group. Ann Intern Med. 1997 Aug 15;127(4):267-74. doi: 10.7326/0003-4819-127-4-199708150-00002. PMID 9265425
- [Background] Rupp ME, Lisco SJ, Lipsett PA, Perl TM, Keating K, Civetta JM, Mermel LA, Lee D, Dellinger EP, Donahoe M, Giles D, Pfaller MA, Maki DG, Sherertz R. Effect of a second-generation venous catheter impregnated with chlorhexidine and silver sulfadiazine on central catheter-related infections: a randomized, controlled trial. Ann Intern Med. 2005 Oct 18;143(8):570-80. doi: 10.7326/0003-4819-143-8-200510180-00007. PMID 16230723
- [Background] Gong P, Li H, He X, et al. Preparation and antibacterial activity of Fe3O4@Ag nanoparticles. Nanotechnology 2007; 18: 604-11
- [Background] Shrivastava S, Bera T, Roy A, Singh G, Ramachandrarao P, Dash D. Retracted: Characterization of enhanced antibacterial effects of novel silver nanoparticles. Nanotechnology. 2007 May 4;18(22). doi: 10.1088/0957-4484/18/22/225103. PMID 37016550
- [Background] Samuel U, Guggenbichler JP. Prevention of catheter-related infections: the potential of a new nano-silver impregnated catheter. Int J Antimicrob Agents. 2004 Mar;23 Suppl 1:S75-8. doi: 10.1016/j.ijantimicag.2003.12.004. PMID 15037331
- [Background] Hsu SH, Tseng HJ, Lin YC. The biocompatibility and antibacterial properties of waterborne polyurethane-silver nanocomposites. Biomaterials. 2010 Sep;31(26):6796-808. doi: 10.1016/j.biomaterials.2010.05.015. Epub 2010 Jun 12. PMID 20542329
- [Background] Lai NM, Chaiyakunapruk N, Lai NA, O'Riordan E, Pau WS, Saint S. Catheter impregnation, coating or bonding for reducing central venous catheter-related infections in adults. Cochrane Database Syst Rev. 2013 Jun 6;(6):CD007878. doi: 10.1002/14651858.CD007878.pub2. PMID 23740696
- [Background] Campisi C, Biffi R, Pittiruti M. Catheter-related venous thrombosis: the development of a nationwide consensus paper in Italy. J AssocVasc Access 2007; 12: 38-46
- [Background] Cortelezzi A, Moia M, Falanga A, Pogliani EM, Agnelli G, Bonizzoni E, Gussoni G, Barbui T, Mannucci PM; CATHEM Study Group. Incidence of thrombotic complications in patients with haematological malignancies with central venous catheters: a prospective multicentre study. Br J Haematol. 2005 Jun;129(6):811-7. doi: 10.1111/j.1365-2141.2005.05529.x. PMID 15953009
- [Background] Kucher N. Clinical practice. Deep-vein thrombosis of the upper extremities. N Engl J Med. 2011 Mar 3;364(9):861-9. doi: 10.1056/NEJMcp1008740. No abstract available. PMID 21366477
- [Background] Monreal M, Raventos A, Lerma R, Ruiz J, Lafoz E, Alastrue A, Llamazares JF. Pulmonary embolism in patients with upper extremity DVT associated to venous central lines--a prospective study. Thromb Haemost. 1994 Oct;72(4):548-50. PMID 7878630
- [Background] Kearon C, Akl EA, Comerota AJ, Prandoni P, Bounameaux H, Goldhaber SZ, Nelson ME, Wells PS, Gould MK, Dentali F, Crowther M, Kahn SR. Antithrombotic therapy for VTE disease: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e419S-e496S. doi: 10.1378/chest.11-2301. PMID 22315268
- [Background] Mehall JR, Saltzman DA, Jackson RJ, Smith SD. Fibrin sheath enhances central venous catheter infection. Crit Care Med. 2002 Apr;30(4):908-12. doi: 10.1097/00003246-200204000-00033. PMID 11940768
- [Background] Raad II, Luna M, Khalil SA, Costerton JW, Lam C, Bodey GP. The relationship between the thrombotic and infectious complications of central venous catheters. JAMA. 1994 Apr 6;271(13):1014-6. PMID 8139059
- [Background] Pierce CM, Wade A, Mok Q. Heparin-bonded central venous lines reduce thrombotic and infective complications in critically ill children. Intensive Care Med. 2000 Jul;26(7):967-72. doi: 10.1007/s001340051289. PMID 10990114
- [Derived] Wu M, Chen Y, Du B, Kang Y. Study protocol for a multicentre, randomised, controlled trial to assess the effectiveness of antimicrobial central venous catheters versus ordinary central venous catheters at reducing catheter related infections in critically ill Chinese patients. BMJ Open. 2017 Dec 29;7(12):e016564. doi: 10.1136/bmjopen-2017-016564. PMID 29289933